CLINICAL TRIAL: NCT03195491
Title: An Open Label, Safety Study of Participants With Non-Small Cell Lung Cancer Receiving Second-Line Nivolumab Monotherapy in Asia
Brief Title: A Study of Non-Small Cell Lung Cancer (NSCLC) Patients Receiving Second-Line Nivolumab Monotherapy in Asia
Acronym: CheckMate870
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA209-870
Record Dates: First submitted 2017-06-20; First posted 2017-06-22 (Actual); Results first posted 2024-07-18 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-01

CONDITIONS: Lung Cancer; Non-Small Cell Lung Cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Monotherapy (Experimental): Nivolumab administered every two weeks
  Interventions: Biological: Nivolumab

INTERVENTIONS:
Biological: Nivolumab — Intravenous infusion administered over 30 minutes at 240 mg
  Other Names: Opdivo; BMS-936558

SUMMARY:
The purpose of this study is to investigate the safety of patients in Asia with Non-Small Cell Lung Cancer (NSCLC)who are treated with Nivolumab monotherapy as a second line or third line treatment.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Advanced metastatic stage IIIB/IV NSCLC (Nonsquamous and squamous)
* 1 to 2 prior systemic therapies
* Eastern Cooperative Oncology Group (ECOG) Performance Status of less than or equal to 1
* Participants must have measurable disease by computed tomography (CT) or magnetic resonance imaging (MRI)
* Prior radiotherapy or radiosurgery must have been completed at least 2 weeks prior to starting study treatment

Exclusion Criteria:

* Women with a positive pregnancy test at enrollment or prior to administration of study medication
* Participants with active central nervous system metastases
* Participants with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of first dose of study drug
* Participants with previous malignancies are excluded unless a complete remission was achieved at least 2 years prior to study entry AND no additional therapy is required or anticipated to be required during the study period
* Participants with carcinomatous meningitis

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2017-12-25 (Actual); Primary Completion 2021-06-08 (Actual); Study Completion 2021-06-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (21):
- China (19):
  - Local Institution, Beijing, Beijing Municipality
  - Local Institution, Fuzhou, Fujian
  - Local Institution, Guangzhou, Guangdong
  - Local Institution, Beijingcun, Hebei
  - Local Institution, Harbin, Heilongjiang
  - Local Institution, Zhengzhou, Henan
  - Local Institution, Wuhan, Hubei
  - Local Institution - 0017, Changsha, Hunan
  - Local Institution, Nanjing, Jiangsu
  - Local Institution, Changchun, Jilin
  - Local Institution, Xi'an, Shan3xi
  - Local Institution, Jinan, Shandong
  - Local Institution, Shanghai, Shanghai Municipality
  - Local Institution, Tianjin, Tianjin Municipality
  - Local Institution, Ürümqi, Xinjiang
  - Local Institution, Hangzhou, Zhejiang
  - Local Institution, Guangzhou
  - Local Institution, Shanghai
  - Local Institution, Shenyang
- Thailand (2):
  - Local Institution, Bangkok
  - Local Institution, Khon Kaen

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Groups:
- Non-HBV Participants: Non-Hepatitis B Virus (HBV) participants who received Nivolumab 240 mg monotherapy/30 minute IV infusion every 2 weeks. Treatment will be given up to 24 months in the absence of disease progression or unacceptable toxicity. Treatment with nivolumab could be reinitiated as per the initial schedule for subsequent disease progression and administered for up to 1 additional year.
- HBV Participants: Hepatitis B Virus (HBV) participants who received Nivolumab 240 mg monotherapy/30 minute IV infusion every 2 weeks. Treatment will be given up to 24 months in the absence of disease progression or unacceptable toxicity. Treatment with nivolumab could be reinitiated as per the initial schedule for subsequent disease progression and administered for up to 1 additional year.
Period: Overall Study
Arm/Group | Non-HBV Participants | HBV Participants
Started | 383 | 17
Completed | 36 | 2
Not Completed | 347 | 15
Not completed — Study drug toxicity | 25 | 3
Not completed — Maximum clinical benefit | 5 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Death | 3 | 0
Not completed — Adverse event unrelated to study drug | 19 | 2
Not completed — Disease progression | 266 | 8
Not completed — Other reasons | 10 | 0
Not completed — Participant withdrew consent | 8 | 1
Not completed — Participant no longer meets study criteria | 0 | 1
Not completed — Participant request to discontinue study treatment | 10 | 0

BASELINE CHARACTERISTICS:
Population: All treated participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Non-HBV Participants | HBV Participants | Total
Number analyzed (Participants) | 383 | 17 | 400
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.6 (8.72) | 59.1 (7.86) | 60.5 (8.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82 | 4 | 86
  Male | 301 | 13 | 314
Race/Ethnicity, Customized [Number; unit: Participants]
  Chinese | 377 | 17 | 394
  Asian Other | 6 | 0 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Non-HBV Participants Experiencing High Grade Treatment-Related Select Adverse Events
Description: Number of non-HBV participants experiencing high grade (combined CTCAE v4 Grade 3-4 and Grade 5) treatment-related select adverse events in non-HBV infected participants. To evaluate safety and tolerability in non-HBV infected participants with advanced or metastatic non-small cell lung cancer (NSCLC) who have progressed during or after one prior systemic therapy and are treated with nivolumab monotherapy with an infusion duration of 30 minutes. Adverse events are graded on a scale from 1 to 5, with Grade 1 being mild and asymptomatic; Grade 2 is moderate requiring minimal, local or noninvasive intervention; Grade 3 is severe or medically significant but not immediately life-threatening; Grade 4 events are usually severe enough to require hospitalization; Grade 5 events are fatal.
Time Frame: From first dose up to 100 days post dose, up to approximately 36 months
Population: All treated non-HBV infected participants
Measure: Count of Participants; unit: Participants
Arm/Group | Non-HBV Participants
Number analyzed (Participants) | 383
Participants
  Gastrointestinal Adverse | 2
  Hepatic Adverse Event | 8
  Pulmonary Adverse Event | 5
  Renal Adverse Event | 2
  Skin Adverse Event | 7

2. Secondary Outcome: Number of HBV Participants Experiencing High Grade Treatment-Related Select Adverse Events
Description: Number of HBV participants experiencing high grade (combined CTCAE v4 Grade 3-4 and Grade 5) treatment-related select adverse events in HBV participants. Adverse events are graded on a scale from 1 to 5, with Grade 1 being mild and asymptomatic; Grade 2 is moderate requiring minimal, local or noninvasive intervention; Grade 3 is severe or medically significant but not immediately life-threatening; Grade 4 events are usually severe enough to require hospitalization; Grade 5 events are fatal.
Time Frame: From first dose up to 100 days post dose, up to approximately 36 months
Population: All treated HBV infected participants
Measure: Count of Participants; unit: Participants
Arm/Group | HBV Participants
Number analyzed (Participants) | 17
Participants
  Gastrointestinal Adverse Event | 0
  Hepatic Adverse Event | 0
  Pulmonary Adverse Event | 0
  Renal Adverse Event | 0
  Skin Adverse Reaction | 1

3. Secondary Outcome: Number of Participants Experiencing Adverse Events (AEs)
Description: An Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a pre-existing medical condition in a clinical investigation participant administered study treatment and that does not necessarily have a causal relationship with this treatment. Adverse events are graded on a scale from 1 to 5, with Grade 1 being mild and asymptomatic; Grade 2 is moderate requiring minimal, local or noninvasive intervention; Grade 3 is severe or medically significant but not immediately life-threatening; Grade 4 events are usually severe enough to require hospitalization; Grade 5 events are fatal.
Time Frame: From first dose up to 100 days post dose, up to approximately 36 months
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Non-HBV Participants | HBV Participants
Number analyzed (Participants) | 383 | 17
Participants | 375 | 17

4. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) is defined as the time from the first dosing date to the date of death. Participants without documentation of death will be recorded on the last date the participant was known to be alive. Tumor PD-L1 protein expression was measured by immunohistochemistry (IHC).
Time Frame: From the first dose up to the date of death. Participants without documentation of death will be censored on the late date known to be alive, up to approximately 32 months
Population: This is a single arm trial with two enrollment cohorts, HPV positive and HPV negative. All participants received the same treatment. Due to the small number of participants in the HPV cohorts, it is not meaningful to perform additional subgroup analysis. For example, there were only 17 participants in the HPV positive cohort, which is less than 5% (17/400 = 4.25%) from the overall. Therefore, all additional efficacy subgroup analysis was performed based on all treated participants.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- All Treated Participants: All treated participants who received Nivolumab 240 mg monotherapy/30 minute IV infusion every 2 weeks. Treatment will be given up to 24 months in the absence of disease progression or unacceptable toxicity. Treatment with nivolumab could be reinitiated as per the initial schedule for subsequent disease progression and administered for up to 1 additional year.
Arm/Group | Non-HBV Participants | HBV Participants | All Treated Participants
Number analyzed (Participants) | 383 | 17 | 400
Months
  All treated participants | 14.16 [12.25 to 18.07] | 22.31 [10.02 to NA] — Upper limit not calculated due to insufficient number of events. | 14.65 [12.32 to 18.10]
  PD-L1 < 1%: number analyzed (Participants) | 0 | 0 | 174
  PD-L1 < 1% |  |  | 13.31 [10.87 to 17.71]
  PD-L1 ≥ 1%: number analyzed (Participants) | 0 | 0 | 168
  PD-L1 ≥ 1% |  |  | 19.25 [12.94 to 23.46]
  PD-L1 < 5%: number analyzed (Participants) | 0 | 0 | 205
  PD-L1 < 5% |  |  | 14.65 [11.63 to 18.10]
  PD-L1 ≥ 5%: number analyzed (Participants) | 0 | 0 | 137
  PD-L1 ≥ 5% |  |  | 18.37 [11.70 to 22.77]
  PD-L1 < 10%: number analyzed (Participants) | 0 | 0 | 222
  PD-L1 < 10% |  |  | 14.72 [12.35 to 18.76]
  PD-L1 ≥ 10%: number analyzed (Participants) | 0 | 0 | 120
  PD-L1 ≥ 10% |  |  | 17.68 [10.78 to 21.03]
  PD-L1 < 50%: number analyzed (Participants) | 0 | 0 | 272
  PD-L1 < 50% |  |  | 16.23 [12.52 to 18.86]
  PD-L1 ≥ 50%: number analyzed (Participants) | 0 | 0 | 70
  PD-L1 ≥ 50% |  |  | 14.75 [10.68 to 29.04]
  PD-L1 Not Reportable: number analyzed (Participants) | 0 | 0 | 58
  PD-L1 Not Reportable |  |  | 11.99 [9.17 to 19.19]
  Squamous Tumor Histology: number analyzed (Participants) | 0 | 0 | 136
  Squamous Tumor Histology |  |  | 13.80 [10.78 to 18.37]
  Non-squamous Tumor Histology: number analyzed (Participants) | 0 | 0 | 264
  Non-squamous Tumor Histology |  |  | 14.75 [11.70 to 19.32]
  EGFR Mutation Positive: number analyzed (Participants) | 0 | 0 | 34
  EGFR Mutation Positive |  |  | 19.32 [11.24 to 31.74]
  ALK translocation positive: number analyzed (Participants) | 0 | 0 | 10
  ALK translocation positive |  |  | 16.48 [1.28 to NA] — Upper limit not reached due to insufficient number of events.

5. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS is the time from first dose to the first documented tumor progression (per RECIST 1.1) or death due to any cause. Participants who die without a reported prior progression are considered to have progressed on their death date. Participants who did not progress or die will be documented on the date of their last evaluable tumor assessment. Participants who did not have any on study tumor assessments and did not die will be documented on their first dose date. Participants who started any subsequent anti-cancer therapy without a prior reported progression will be documented at the last evaluable tumor assessment prior to initiation of the subsequent anti-cancer therapy. Tumor PD-L1 protein expression was measured by immunohistochemistry (IHC). Per RECIST v1.0 for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: From the first dose up to the date of the first documented tumor progression (per RECIST 1.1) or death due to any cause, up to approximately 30 months
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Non-HBV Participants | HBV Participants | All Treated Participants
Number analyzed (Participants) | 383 | 17 | 400
Months
  All treated participants | 3.61 [2.33 to 3.75] | 2.04 [1.64 to 10.22] | 3.61 [2.33 to 3.75]
  PD-L1 < 1%: number analyzed (Participants) | 0 | 0 | 174
  PD-L1 < 1% |  |  | 2.33 [1.94 to 3.68]
  PD-L1 ≥ 1%: number analyzed (Participants) | 0 | 0 | 168
  PD-L1 ≥ 1% |  |  | 4.73 [3.68 to 5.65]
  PD-L1 < 5: number analyzed (Participants) | 0 | 0 | 205
  PD-L1 < 5 |  |  | 2.37 [1.94 to 3.68]
  PD-L1 ≥ 5: number analyzed (Participants) | 0 | 0 | 137
  PD-L1 ≥ 5 |  |  | 5.42 [3.68 to 5.65]
  PD-L1 < 10: number analyzed (Participants) | 0 | 0 | 222
  PD-L1 < 10 |  |  | 2.50 [1.94 to 3.68]
  PD-L1 ≥ 10: number analyzed (Participants) | 0 | 0 | 120
  PD-L1 ≥ 10 |  |  | 5.45 [3.68 to 5.65]
  PD-L1 < 50: number analyzed (Participants) | 0 | 0 | 272
  PD-L1 < 50 |  |  | 3.58 [2.07 to 3.75]
  PD-L1 ≥ 50: number analyzed (Participants) | 0 | 0 | 70
  PD-L1 ≥ 50 |  |  | 5.55 [2.23 to 7.33]
  EGFR mutation positive: number analyzed (Participants) | 0 | 0 | 34
  EGFR mutation positive |  |  | 1.87 [1.71 to 4.73]
  ALK translocation positive: number analyzed (Participants) | 0 | 0 | 10
  ALK translocation positive |  |  | 1.91 [1.28 to 16.36]
  Squamous subgroup: number analyzed (Participants) | 0 | 0 | 136
  Squamous subgroup |  |  | 3.75 [3.06 to 5.55]
  Non-squamous subgroup: number analyzed (Participants) | 0 | 0 | 264
  Non-squamous subgroup |  |  | 2.79 [1.94 to 3.68]

6. Secondary Outcome: Number of Participants Experiencing Laboratory Abnormalities in Specific Liver Tests
Description: Number of Participants experiencing laboratory abnormalities are defined as on-study lab parameters summarized by using the worst grade per NCI CTCAE v.4 criteria
Time Frame: From first dose up to 100 days post last dose, up to approximately 36 months
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Non-HBV Participants | HBV Participants
Number analyzed (Participants) | 383 | 17
Participants
  ALT OR AST > 3XULN | 16 | 1
  ALT OR AST > 5XULN | 5 | 0
  ALT OR AST > 10XULN | 4 | 0
  ALT OR AST > 20XULN | 2 | 0
  TOTAL BILIRUBIN > 2XULN | 4 | 0
  CONCURRENT ALT OR AST ELEVATION > 3XULN WITH TOTAL BILIRUBIN > 2XULN WITHIN ONE DAY | 0 | 0
  CONCURRENT ALT OR AST ELEVATION > 3XULN WITH TOTAL BILIRUBIN > 2XULN WITHIN 30 DAY | 0 | 0

7. Secondary Outcome: Number of Participants Experiencing Serious Adverse Events (SAEs)
Description: Number of Participants experiencing SAEs are tabulated using worst grade per NCI CTCAE v.4 criteria by system organ class and MedDRA preferred term.
Time Frame: From first dose to 100 days post last dose, up to 36 months
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Non-HBV Participants | HBV Participants
Number analyzed (Participants) | 383 | 17
Participants | 157 | 12

8. Secondary Outcome: Objective Response Rate
Description: Objective Response Rate (ORR) is defined as the percentage of all treated subjects whose best overall response (BOR) from baseline is either a CR or PR per RECIST 1.1 criteria. BOR is determined by the best response designation recorded between the first dose date and the date of objectively documented progression or the date of subsequent anti-cancer therapy, whichever occurs first. For subjects without documented progression or subsequent anticancer therapy, all available response designations will contribute to the BOR determination. For subjects who continue nivolumab beyond progression, the BOR should be determined based on response designations recorded at the time of the initial RECIST 1.1 defined progression.
Time Frame: From the first dose date up to the date of objectively documented progression or the date of subsequent anti-cancer therapy, whichever occurs first. Up to approximately 36 months
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Non-HBV Participants | HBV Participants | All Treated Participants
Number analyzed (Participants) | 383 | 17 | 400
Percentage of participants
  All treated participants | 14.88 [11.47 to 18.85] | 17.65 [3.80 to 43.43] | 15.00 [11.65 to 18.88]
  Squamous tumor histology: number analyzed (Participants) | 0 | 0 | 136
  Squamous tumor histology |  |  | 18.38 [12.26 to 25.93]
  Non-squamous tumor histology: number analyzed (Participants) | 0 | 0 | 264
  Non-squamous tumor histology |  |  | 13.26 [9.41 to 17.95]
  PD-L1 < 1%: number analyzed (Participants) | 0 | 0 | 174
  PD-L1 < 1% |  |  | 6.32 [3.20 to 11.03]
  PD-L1 ≥ 1%: number analyzed (Participants) | 0 | 0 | 168
  PD-L1 ≥ 1% |  |  | 25.60 [19.18 to 32.89]
  PD-L1 < 5%: number analyzed (Participants) | 0 | 0 | 205
  PD-L1 < 5% |  |  | 8.78 [5.29 to 13.52]
  PD-L1 ≥ 5%: number analyzed (Participants) | 0 | 0 | 137
  PD-L1 ≥ 5% |  |  | 26.28 [19.13 to 34.48]
  PD-L1 < 10%: number analyzed (Participants) | 0 | 0 | 222
  PD-L1 < 10% |  |  | 10.81 [7.05 to 15.66]
  PD-L1 ≥ 10%: number analyzed (Participants) | 0 | 0 | 120
  PD-L1 ≥ 10% |  |  | 25.00 [17.55 to 33.73]
  PD-L1 < 50%: number analyzed (Participants) | 0 | 0 | 272
  PD-L1 < 50% |  |  | 11.76 [8.19 to 16.20]
  PD-L1 ≥ 50%: number analyzed (Participants) | 0 | 0 | 70
  PD-L1 ≥ 50% |  |  | 31.43 [20.85 to 43.63]
  EGFR mutation positive: number analyzed (Participants) | 0 | 0 | 34
  EGFR mutation positive |  |  | 17.65 [6.76 to 34.53]
  ALK translocation positive: number analyzed (Participants) | 0 | 0 | 10
  ALK translocation positive |  |  | 10.00 [0.25 to 44.50]

9. Secondary Outcome: Duration of Tumor Response
Description: Duration of Response (DOR) is defined as the time between the date of first confirmed response to the date of the first documented tumor progression (per RECIST 1.1) or death due to any cause. Participants who neither progress nor die will be documented on the date of their last assessment. The censoring algorithm for DOR will be the same as used for PFS definition. This endpoint will only be evaluated for participants with the best overall response of complete response or partial response.
Time Frame: From the date of first confirmed response to the date of the first documented tumor progression, up to approximately 30 months
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | HBV Participants | Non-HBV Participants | All Treated Participants
Number analyzed (Participants) | 3 | 57 | 60
Months
  All treated participants | NA [8.15 to NA] — Median and upper limit not reached due to insufficient number of events. | 19.38 [11.04 to 24.97] | 19.38 [11.04 to 24.97]
  Squamous tumor histology: number analyzed (Participants) | 0 | 0 | 25
  Squamous tumor histology |  |  | 12.62 [8.11 to 25.33]
  Non-squamous tumor histology: number analyzed (Participants) | 0 | 0 | 34
  Non-squamous tumor histology |  |  | 19.61 [9.49 to 27.60]
  PD-L1 < 1%: number analyzed (Participants) | 0 | 0 | 11
  PD-L1 < 1% |  |  | 19.38 [8.11 to 24.97]
  PD-L1 ≥ 1%: number analyzed (Participants) | 0 | 0 | 42
  PD-L1 ≥ 1% |  |  | 16.11 [9.43 to 27.60]
  PD-L1 < 5%: number analyzed (Participants) | 0 | 0 | 17
  PD-L1 < 5% |  |  | 19.38 [8.11 to 24.97]
  PD-L1 ≥ 5%: number analyzed (Participants) | 0 | 0 | 36
  PD-L1 ≥ 5% |  |  | 19.61 [9.33 to 29.70]
  PD-L1 < 10%: number analyzed (Participants) | 0 | 0 | 23
  PD-L1 < 10% |  |  | 12.06 [8.11 to 24.97]
  PD-L1 ≥ 10%: number analyzed (Participants) | 0 | 0 | 30
  PD-L1 ≥ 10% |  |  | 21.13 [9.43 to NA] — Upper limit not reached due to insufficient number of events.
  PD-L1 < 50%: number analyzed (Participants) | 0 | 0 | 31
  PD-L1 < 50% |  |  | 12.06 [8.15 to 24.97]
  PD-L1 ≥ 50%: number analyzed (Participants) | 0 | 0 | 22
  PD-L1 ≥ 50% |  |  | 21.49 [9.30 to NA] — Upper limit not reached due to insufficient number of events.
  EGFR mutation positive: number analyzed (Participants) | 0 | 0 | 6
  EGFR mutation positive |  |  | 12.57 [5.59 to NA] — Upper limit not reached due to insufficient number of events.
  ALK translocation positive: number analyzed (Participants) | 0 | 0 | 1
  ALK translocation positive |  |  | 19.42 [NA to NA] — Lower and upper limits not reached due to insufficient number of events.

10. Secondary Outcome: Number of Participants Experiencing Laboratory Abnormalities in Specific Thyroid Tests
Description: as for outcome 6
Time Frame: From randomization to 100 days post last dose, up to 36 months
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Non-HBV Participants | HBV Participants
Number analyzed (Participants) | 383 | 17
Participants
  TSH > ULN | 87 | 1
  TSH > ULN WITH TSH <= ULN AT BASELINE | 63 | 0
  TSH > ULN WITH AT LEAST ONE FT3/FT4 TEST VALUE < LLN | 36 | 1
  TSH > ULN WITH ALL OTHER FT3/FT4 TEST VALUES >= LLN | 52 | 0
  TSH > ULN WITH FT3/FT4 TEST MISSING | 74 | 1
  TSH < LLN | 66 | 3
  TSH < LLN WITH TSH >= LLN AT BASELINE | 56 | 3
  TSH < LLN WITH AT LEAST ONE FT3/FT4 TEST VALUE > ULN | 34 | 1
  TSH < LLN WITH ALL OTHER FT3/FT4 TEST VALUES <= ULN | 32 | 2
  TSH < LLN WITH FT3/FT4 TEST MISSING | 43 | 2

11. Secondary Outcome: Time to Treatment Failure (TTF)
Description: Time to Treatment Failure is defined as the minimum of the time from treatment assignment to disease progression (determined by investigator assessments using RECIST 1.1), death or last dose date if a participant progressed, died or discontinued from treatment for any reasons other than "maximum clinical benefit" and "administrative reasons by sponsor". TTF is censored at the last dose date for participants who continued on treatment without progression (per RECIST 1.1) or death at the time of the database lock. Tumor PD-L1 protein expression was measured by immunohistochemistry (IHC).
Time Frame: From treatment assignment to disease progression, death or last dose date, up to approximately 16 months
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Non-HBV Participants | HBV Participants | All Treated Participants
Number analyzed (Participants) | 383 | 17 | 400
Months
  All treated participants | 2.23 [1.94 to 3.52] | 1.97 [1.41 to 10.22] | 2.10 [1.94 to 3.52]
  Squamous Tumor Histology: number analyzed (Participants) | 0 | 0 | 136
  Squamous Tumor Histology |  |  | 3.68 [2.10 to 5.45]
  Non-Squamous Tumor Histology: number analyzed (Participants) | 0 | 0 | 264
  Non-Squamous Tumor Histology |  |  | 1.94 [1.87 to 2.50]
  EGFR Mutation Positive: number analyzed (Participants) | 0 | 0 | 34
  EGFR Mutation Positive |  |  | 1.86 [1.68 to 3.65]
  ALK Translocation Positive: number analyzed (Participants) | 0 | 0 | 10
  ALK Translocation Positive |  |  | 1.91 [1.28 to 16.36]
  PD-L1 < 1%: number analyzed (Participants) | 0 | 0 | 174
  PD-L1 < 1% |  |  | 1.97 [1.87 to 2.92]
  PD-L1 ≥ 1%: number analyzed (Participants) | 0 | 0 | 168
  PD-L1 ≥ 1% |  |  | 3.68 [2.17 to 5.55]
  PD-L1 < 5%: number analyzed (Participants) | 0 | 0 | 205
  PD-L1 < 5% |  |  | 1.97 [1.87 to 3.06]
  PD-L1 ≥ 5%: number analyzed (Participants) | 0 | 0 | 137
  PD-L1 ≥ 5% |  |  | 3.68 [2.23 to 5.55]
  PD-L1 < 10%: number analyzed (Participants) | 0 | 0 | 222
  PD-L1 < 10% |  |  | 1.97 [1.87 to 3.09]
  PD-L1 ≥ 10%: number analyzed (Participants) | 0 | 0 | 120
  PD-L1 ≥ 10% |  |  | 3.75 [2.23 to 5.55]
  PD-L1 < 50%: number analyzed (Participants) | 0 | 0 | 272
  PD-L1 < 50% |  |  | 2.14 [1.91 to 3.58]
  PD-L1 ≥ 50%: number analyzed (Participants) | 0 | 0 | 70
  PD-L1 ≥ 50% |  |  | 4.11 [2.00 to 6.01]

ADVERSE EVENTS:
Time Frame: All-cause mortality was assessed from date of first dose to study completion (up to approximately 41 months). Serious Adverse events and other adverse events were assessed from date of first dose to 100 days following date of last dose (up to approximately 36 months).
Groups:
- TOTAL: All treated participants who received Nivolumab 240 mg monotherapy/30 minute IV infusion every 2 weeks. Treatment will be given up to 24 months in the absence of disease progression or unacceptable toxicity. Treatment with nivolumab could be reinitiated as per the initial schedule for subsequent disease progression and administered for up to 1 additional year.
Arm/Group | Non-HBV Participants | HBV Participants | TOTAL
All-Cause Mortality (participants affected / at risk) | 270/383 | 9/17 | 279/400
Serious Adverse Events (participants affected / at risk) | 157/383 | 12/17 | 169/400
Other Adverse Events (participants affected / at risk) | 359/383 | 17/17 | 376/400
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Non-HBV Participants (N=383) | HBV Participants (N=17) | TOTAL (N=400)
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 2
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 1
Arrhythmia (Cardiac disorders) | 1 | 0 | 1
Cardiac failure (Cardiac disorders) | 2 | 0 | 2
Immune-mediated myocarditis (Cardiac disorders) | 1 | 0 | 1
Myocarditis (Cardiac disorders) | 1 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 0 | 1
Ventricular fibrillation (Cardiac disorders) | 1 | 0 | 1
Hypothyroidism (Endocrine disorders) | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1
Ascites (Gastrointestinal disorders) | 2 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 3 | 0 | 3
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 0 | 1
Oesophageal obstruction (Gastrointestinal disorders) | 2 | 0 | 2
Death (General disorders) | 2 | 1 | 3
Malaise (General disorders) | 2 | 0 | 2
Multiple organ dysfunction syndrome (General disorders) | 1 | 0 | 1
Oedema (General disorders) | 1 | 0 | 1
Pyrexia (General disorders) | 2 | 1 | 3
Sudden death (General disorders) | 2 | 0 | 2
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 5 | 0 | 5
Liver injury (Hepatobiliary disorders) | 2 | 0 | 2
Contrast media allergy (Immune system disorders) | 1 | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0 | 1
Bacteraemia (Infections and infestations) | 1 | 0 | 1
Endophthalmitis (Infections and infestations) | 1 | 0 | 1
Lymphangitis (Infections and infestations) | 1 | 0 | 1
Pneumonia (Infections and infestations) | 29 | 4 | 33
Pulmonary tuberculosis (Infections and infestations) | 1 | 0 | 1
Septic shock (Infections and infestations) | 1 | 0 | 1
Soft tissue infection (Infections and infestations) | 1 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 4 | 0 | 4
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Blood creatinine increased (Investigations) | 2 | 0 | 2
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 1
Platelet count decreased (Investigations) | 3 | 0 | 3
Troponin I increased (Investigations) | 1 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0 | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 0 | 2
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 1 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 0 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Benign neoplasm of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 19 | 0 | 19
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1 | 4
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Altered state of consciousness (Nervous system disorders) | 1 | 0 | 1
Ataxia (Nervous system disorders) | 1 | 0 | 1
Cerebral infarction (Nervous system disorders) | 4 | 0 | 4
Dizziness (Nervous system disorders) | 1 | 0 | 1
Epilepsy (Nervous system disorders) | 1 | 0 | 1
Lacunar infarction (Nervous system disorders) | 1 | 0 | 1
Spinal cord compression (Nervous system disorders) | 0 | 1 | 1
Vascular headache (Nervous system disorders) | 1 | 0 | 1
Completed suicide (Psychiatric disorders) | 1 | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0 | 1
Proteinuria (Renal and urinary disorders) | 1 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Choking (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 2 | 8
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 12 | 0 | 12
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 8 | 1 | 9
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 10 | 0 | 10
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 4
Tracheal fistula (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Hypotension (Vascular disorders) | 1 | 0 | 1
Superior vena cava syndrome (Vascular disorders) | 1 | 0 | 1
Venous thrombosis limb (Vascular disorders) | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Non-HBV Participants (N=383) | HBV Participants (N=17) | TOTAL (N=400)
Anaemia (Blood and lymphatic system disorders) | 155 | 7 | 162
Leukocytosis (Blood and lymphatic system disorders) | 21 | 4 | 25
Hyperthyroidism (Endocrine disorders) | 28 | 0 | 28
Hypothyroidism (Endocrine disorders) | 48 | 1 | 49
Constipation (Gastrointestinal disorders) | 39 | 3 | 42
Diarrhoea (Gastrointestinal disorders) | 28 | 2 | 30
Nausea (Gastrointestinal disorders) | 41 | 1 | 42
Vomiting (Gastrointestinal disorders) | 26 | 2 | 28
Asthenia (General disorders) | 33 | 3 | 36
Chest discomfort (General disorders) | 18 | 3 | 21
Fatigue (General disorders) | 60 | 2 | 62
Malaise (General disorders) | 50 | 2 | 52
Non-cardiac chest pain (General disorders) | 26 | 1 | 27
Pyrexia (General disorders) | 72 | 6 | 78
Pneumonia (Infections and infestations) | 41 | 3 | 44
Upper respiratory tract infection (Infections and infestations) | 37 | 3 | 40
Alanine aminotransferase increased (Investigations) | 62 | 4 | 66
Aspartate aminotransferase increased (Investigations) | 59 | 5 | 64
Blood alkaline phosphatase increased (Investigations) | 21 | 0 | 21
Blood bilirubin increased (Investigations) | 22 | 1 | 23
Blood creatinine increased (Investigations) | 23 | 0 | 23
Blood lactate dehydrogenase increased (Investigations) | 25 | 1 | 26
Blood urea increased (Investigations) | 21 | 0 | 21
Gamma-glutamyltransferase increased (Investigations) | 30 | 0 | 30
Neutrophil count decreased (Investigations) | 21 | 0 | 21
Platelet count decreased (Investigations) | 21 | 1 | 22
Weight decreased (Investigations) | 66 | 1 | 67
Weight increased (Investigations) | 21 | 2 | 23
Decreased appetite (Metabolism and nutrition disorders) | 94 | 2 | 96
Hyperglycaemia (Metabolism and nutrition disorders) | 32 | 1 | 33
Hypoalbuminaemia (Metabolism and nutrition disorders) | 46 | 3 | 49
Hypocalcaemia (Metabolism and nutrition disorders) | 21 | 1 | 22
Hypokalaemia (Metabolism and nutrition disorders) | 41 | 2 | 43
Hyponatraemia (Metabolism and nutrition disorders) | 52 | 6 | 58
Hypoproteinaemia (Metabolism and nutrition disorders) | 26 | 1 | 27
Arthralgia (Musculoskeletal and connective tissue disorders) | 29 | 1 | 30
Back pain (Musculoskeletal and connective tissue disorders) | 34 | 0 | 34
Headache (Nervous system disorders) | 20 | 1 | 21
Insomnia (Psychiatric disorders) | 25 | 1 | 26
Cough (Respiratory, thoracic and mediastinal disorders) | 85 | 7 | 92
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 48 | 3 | 51
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 37 | 0 | 37
Productive cough (Respiratory, thoracic and mediastinal disorders) | 49 | 3 | 52
Rash (Skin and subcutaneous tissue disorders) | 50 | 3 | 53
Granulocytosis (Blood and lymphatic system disorders) | 1 | 1 | 2
Leukopenia (Blood and lymphatic system disorders) | 9 | 1 | 10
Neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 2
Arrhythmia (Cardiac disorders) | 4 | 1 | 5
Atrial fibrillation (Cardiac disorders) | 4 | 1 | 5
Cardiac failure (Cardiac disorders) | 1 | 1 | 2
Pericardial effusion (Cardiac disorders) | 2 | 1 | 3
Supraventricular tachycardia (Cardiac disorders) | 6 | 1 | 7
Dry eye (Eye disorders) | 1 | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 10 | 1 | 11
Abdominal pain lower (Gastrointestinal disorders) | 3 | 1 | 4
Abdominal pain upper (Gastrointestinal disorders) | 9 | 1 | 10
Chronic gastritis (Gastrointestinal disorders) | 2 | 1 | 3
Gingival pain (Gastrointestinal disorders) | 2 | 1 | 3
Toothache (Gastrointestinal disorders) | 9 | 1 | 10
Oedema peripheral (General disorders) | 17 | 1 | 18
Pain (General disorders) | 6 | 1 | 7
Liver injury (Hepatobiliary disorders) | 5 | 2 | 7
Anaphylactic reaction (Immune system disorders) | 0 | 1 | 1
Bronchitis (Infections and infestations) | 4 | 1 | 5
Hepatitis C (Infections and infestations) | 0 | 1 | 1
Paronychia (Infections and infestations) | 1 | 1 | 2
Pharyngitis (Infections and infestations) | 0 | 1 | 1
Tooth infection (Infections and infestations) | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 11 | 1 | 12
Eye injury (Injury, poisoning and procedural complications) | 0 | 1 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 1
Blood albumin decreased (Investigations) | 5 | 2 | 7
Blood glucose increased (Investigations) | 8 | 1 | 9
Blood phosphorus decreased (Investigations) | 4 | 1 | 5
Blood uric acid decreased (Investigations) | 0 | 1 | 1
Blood uric acid increased (Investigations) | 9 | 1 | 10
Brain natriuretic peptide increased (Investigations) | 2 | 1 | 3
C-reactive protein increased (Investigations) | 6 | 1 | 7
Carcinoembryonic antigen increased (Investigations) | 0 | 1 | 1
Gastric pH decreased (Investigations) | 0 | 1 | 1
Haemoglobin decreased (Investigations) | 2 | 1 | 3
Hepatitis B DNA increased (Investigations) | 0 | 1 | 1
Neutrophil count increased (Investigations) | 15 | 4 | 19
Neutrophil percentage increased (Investigations) | 1 | 1 | 2
Procalcitonin increased (Investigations) | 1 | 1 | 2
Red blood cell sedimentation rate increased (Investigations) | 0 | 1 | 1
Tri-iodothyronine free increased (Investigations) | 5 | 1 | 6
Volume blood decreased (Investigations) | 0 | 1 | 1
White blood cell count decreased (Investigations) | 20 | 0 | 20
Acidosis (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 7 | 1 | 8
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 | 1 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 7 | 1 | 8
Hyperuricaemia (Metabolism and nutrition disorders) | 18 | 1 | 19
Hypochloraemia (Metabolism and nutrition disorders) | 15 | 2 | 17
Hypomagnesaemia (Metabolism and nutrition disorders) | 5 | 1 | 6
Hypophosphataemia (Metabolism and nutrition disorders) | 8 | 2 | 10
Tetany (Metabolism and nutrition disorders) | 0 | 1 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 7 | 1 | 8
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 5 | 2 | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 14 | 3 | 17
Dizziness (Nervous system disorders) | 16 | 2 | 18
Neuropathy peripheral (Nervous system disorders) | 1 | 1 | 2
Spinal cord compression (Nervous system disorders) | 1 | 1 | 2
Trigeminal neuralgia (Nervous system disorders) | 0 | 1 | 1
Bronchial haemorrhage (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 4
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 6
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 6 | 1 | 7
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 4
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 3
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 4
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Eczema (Skin and subcutaneous tissue disorders) | 3 | 1 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 16 | 2 | 18
Hypertension (Vascular disorders) | 12 | 2 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Study Protocol (2017-10-25): https://cdn.clinicaltrials.gov/large-docs/91/NCT03195491/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-16): https://cdn.clinicaltrials.gov/large-docs/91/NCT03195491/SAP_001.pdf